CLINICAL TRIAL: NCT04316130
Title: Hospital-home Linkage Short-term Rehabilitation Therapy Using Real-time Interactive Digital Healthcare System in Frozen Shoulder; Randomized Controlled Trial, Assessor Blinding, Multi-center Study
Brief Title: Real-time Interactive Digital Healthcare System in Frozen Shoulder; Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC-2019-05-021
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Range of motion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise using Uincare Homeplus (Experimental): Uincare Homeplus
  Interventions: Device: Uincare Homeplus
- Exercise using brochure (Active Comparator): brochure
  Interventions: Other: Brochure

INTERVENTIONS:
Device: Uincare Homeplus — Interactive digital healthcare system
  Other Names: digital healthcare
  Arms: Exercise using Uincare Homeplus
Other: Brochure — Brochure
  Arms: Exercise using brochure

SUMMARY:
This study aims to examine the effect of hospital-home linkage short-term rehabilitation therapy using real-time interactive digital healthcare system (Uincare Homeplus) in frozen shoulder. This is prospective randomized controlled trial and multi-center study. 100 frozen shoulder who diagnosed with limited range of motion in 2 more plane of flexion, abduction, external rotation of affected shoulder. Shoulder range of motion (ROM), Shoulder Pain and Disability Index (SPADI), pain evaluation with Numeral Rating Scale (NRS), quality of life evaluation with Short Form (SF)-36 Health Survey and EQ-5D-5L, activity daily living (ADL) evaluation with Canadian Occupational Performance Measure (COPM) will be evaluated on enrollment, 4-week, 8-week, 12-weeks, 18-weeks, and 24 weeks after enrollment.

DETAILED DESCRIPTION:
The frozen shoulder is a disease in which severe pain and limited range of motion of the shoulder occur as an inflammatory change occurs in the articular capsular surrounding the shoulder joint. As a result, it has caused limitation in daily life movement.

Uincare Homeplus is software manufactured in Korea, which uses infrared, kinect camera and motion capture technology to track 3D motion of the patients' articulation. Using this technology, the patients can receive feedback of their motion immediately.

The objective of the study is to examine the effect of hospital-home linkage short-term rehabilitation therapy using real-time interactive digital healthcare system (Uincare Homeplus) in frozen shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Limited passive range of motion of the affected shoulder in 2 more plane (flexion < 150˚, abduction <150˚, external rotation < 60˚)

Exclusion Criteria:

* Bilateral frozen shoulder
* Secondary frozen shoulder caused by trauma (shoulder fracture, dislocation), or/and inflammatory disease(rheumatoid arthritis)
* Those unable to perform exercise due to general deconditioning
* Those with communication difficulty

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Range of motion (ROM) in affected shoulder | Enrollment, 4 week, 8 week, 12 week, 18 weeks, 24 weeks
  Evaluation of change of ROM in the affected shoulder from baseline to 12 weeks

SECONDARY OUTCOMES:
Functional outcome in patients with frozen shoulder using Shoulder Pain and Disability Index (SPADI) | Enrollment, 4 week, 8 week, 12 week, 18 weeks, 24 weeks
  Evaluation of shoulder function (pain and disability) using SPADI. Overall total scores range from 0 to 130 with a percentage score of 0 indicating less shoulder disability and 100 indicating more shoulder dysfunction.
Numerical rating scale (NRS) of affected shoulder | Enrollment, 4 week, 8 week, 12 week, 18 weeks, 24 weeks
  Evaluation of pain of the affected shoulder using numerical rating scale (0-10, with score 0 indicating no pain) minimum ~ maximum value: 0 ~ 10, higher scores mean worse outcome.
Quality of life in the patients with frozen shoulder using Short form -36 (SF36) | Enrollment, 4 week, 8 week, 12 week, 18 weeks, 24 weeks
  Evaluation of quality of life using SF36. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Quality of life in the patients with frozen shoulder using EQ-5D-5L | Enrollment, 4 week, 8 week, 12 week, 18 weeks, 24 weeks
  Evaluation of quality of life using EQ-5D-5L. This scale is numbered from -0.066 to 0.904. lower value means the worst quality of life you can imagine.
Activities of Daily Living of the patients with frozen shoulder using Canadian Occupational Performance Measure (COPM) | Enrollment, 4 week, 8 week, 12 week, 18 weeks, 24 weeks
  Evaluation of quality of life using COPM PERFORMANCE and SATISFACTION scores can be generated for up to 5 individual occupational performance problems. Average PERFORMANCE and SATISFACTION scores can be calculated by summing individual problem scores and dividing by the number of problems. Change scores for both PERFORMANCE and SATISFACTION can be calculated after a reassessment interval.

CONTACTS AND LOCATIONS:
Overall Officials: JIHYE HWANG, Professor, Study Chair — Physical & Rehabilitation Medicine Samsung Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Department of rehabilitation, Seoul St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Seoul, Seocho-gu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yeo SM, Lim JY, Kim S, Park HY, Lim JY, Do JG, Lee JI, Hwang JH. Effects of augmented reality-based telerehabilitation in adhesive capsulitis of the shoulder: a randomized controlled trial. Ann Phys Rehabil Med. 2025 Jun;68(5):101956. doi: 10.1016/j.rehab.2025.101956. Epub 2025 Jun 27. PMID 40580799
- [Derived] Yeo SM, Lim JY, Do JG, Lim JY, In Lee J, Hwang JH. Effectiveness of interactive augmented reality-based telerehabilitation in patients with adhesive capsulitis: protocol for a multi-center randomized controlled trial. BMC Musculoskelet Disord. 2021 Apr 26;22(1):386. doi: 10.1186/s12891-021-04261-1. PMID 33902546